CLINICAL TRIAL: NCT06074874
Title: Intestinal Biomarker Analysis After ECP for ICI Colitis
Acronym: IBA_ECP
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Robert Zeiser, Director Division of Tumor immunology, University of Freiburg
Other Study IDs: ICI_colitis_ECP
Record Dates: First submitted 2023-09-28; First posted 2023-10-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Colitis; Immune Checkpoint Inhibitor-Related Colitis
MeSH Terms: conditions — Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — intestinal biopsies and peripheral blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intestinal tissue analysis — Intestinal tissue analysis

SUMMARY:
It was previously shown that ICI-colitis can be treated with extracorporeal photophoresis. Therefore this retrospective analysis is launched to study the chnages of immune cells in the peripheral blood and intestinal tract in an ICI colitis patient cohort. The analysis will include the evaluation of intestinal and peripheral blood biomarkers in patients with ICI colitis receiving ECP as a treatment.

DETAILED DESCRIPTION:
It was previously shown that ICI-colitis can be treated with extracorporeal photophoresis. Therefore this retrospective analysis is launched to study the changes of immune cells in the peripheral blood and intestinal tract in an ICI colitis patient cohort. The analysis will include the evaluation of intestinal and peripheral blood biomarkers in patients with ICI colitis receiving ECP as a treatment.

ELIGIBILITY:
Inclusion Criteria:

* ICI colitis

Exclusion Criteria:

* no informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ICI colitis
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
T cell number and phenotype measurement in the intestinal tract | 6 months
  Analysis of CD3+ T cells by flow cytometry

SECONDARY OUTCOMES:
T cell number measurement by immunohistochemistry | 6 months
  Analysis of CD3+ T cells by immunohistochemistry
Analysis of arginase amounts in the intestinal tract using qPCR | 6 months
  Analysis of arginase mRNA expression by realtime PCR (qRT-PCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Freiburg University Medical Center, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Apostolova P, Unger S, von Bubnoff D, Meiss F, Becher B, Zeiser R. Extracorporeal Photopheresis for Colitis Induced by Checkpoint-Inhibitor Therapy. N Engl J Med. 2020 Jan 16;382(3):294-296. doi: 10.1056/NEJMc1912274. No abstract available. PMID 31940706
- [Result] Maas-Bauer K, Kiote-Schmidt C, Bertz H, Apostolova P, Wasch R, Ihorst G, Finke J, Zeiser R. Ruxolitinib-ECP combination treatment for refractory severe chronic graft-versus-host disease. Bone Marrow Transplant. 2021 Apr;56(4):909-916. doi: 10.1038/s41409-020-01122-8. Epub 2020 Nov 17. PMID 33203951